CLINICAL TRIAL: NCT00672750
Title: A Retrospective Review Of Outcomes Following Laparoscopic Myomectomy
Acronym: retromyo
Status: Terminated | Type: Observational
Why Stopped: did not have resources to continue this study
Sponsor: The Advanced Gynecologic Surgery Institute (Other)
Responsible Party: Principal Investigator, Charles E Miller MD, Principal Investigator, The Advanced Gynecologic Surgery Institute
Other Study IDs: 23597
Record Dates: First submitted 2008-05-01; First posted 2008-05-06 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Laparoscopic Myomectomy
Keywords: laparoscopic; myomectomy; menorrhagia; pelvic pain
MeSH Terms: conditions — Menorrhagia; Pelvic Pain

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- I: Patients of Dr C Miller who have undergone laparoscopic myomectomy from 1999- to present

SUMMARY:
This will be a retrospective review of approximately 900 patients who have undergone laparoscopic myomectomy since 1999. patients will be contacted by phone and surveyed. All patients who have had laparoscopic myomectomy will be included. Only those not wishing to take part in the survey will be excluded. The data will then be compiled for statistical analysis , looking at pain, bleeding and subsequent fertility.

DETAILED DESCRIPTION:
Patients will be called and surveyed using a survey tool. They will be asked about what factors lead them to have surgery and then was their issue resolved after surgery.

ELIGIBILITY:
Inclusion Criteria:

* All patients who are willing to be surveyed

Exclusion Criteria:

* Those patients who are not willing to answer the survey will be excluded

  * Those patients who are unable to be contacted( ie; moved) will be excluded

Ages: 16 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Private patients of Dr Charles Miller who have undergone laparoscopic myomectomy since 1999
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2008-02; Primary Completion 2016-09-16 (Actual); Study Completion 2016-09-16 (Actual)

PRIMARY OUTCOMES:
That patients who had pain prior to laparoscopic myomectomy will have less pain in 75% of the cases | since 1999

SECONDARY OUTCOMES:
That patients who had menorrhagia prior to laparoscopic myomectomy would see a reduction after surgery 75% of the time | since 1999

CONTACTS AND LOCATIONS:
Overall Officials: Charles E Miller, MD, Principal Investigator — Advanced gynecologic surgery institute
Locations (1):
- Advanced Gynecologic Surgery Institute, Naperville, Illinois, United States